CLINICAL TRIAL: NCT02271880
Title: Improving Medication Adherence in ADHD Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was stopped prematurely due to low enrollment.
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH097819
Record Dates: First submitted 2014-09-24; First posted 2014-10-22 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: ADHD
Keywords: Medication nonadherence
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Medication Adherence | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication as usual (Active Comparator): Medication as typically prescribed by physician.
  Interventions: Other: Medication as usual
- Medication as usual + STAR (Active Comparator): Medication as typically prescribed with the addition of the psychosocial intervention to improve medication adherence
  Interventions: Other: Medication as usual; Other: STAR

INTERVENTIONS:
Other: Medication as usual — Physicians will prescribe medication as usual to the adolescent.
Other: STAR — Adolescents and their parents will receive 6 sessions of psychosocial treatment to improve adolescents' motivation to use medication and to develop parent/teen contracting with the goal of setting medication adherence goals.
  Arms: Medication as usual + STAR

SUMMARY:
Investigates whether a family-based intervention for adolescents with Attention Deficit Hyperactivity Disorder (ADHD) will improve adherence to prescribed medication regimen in adolescents with history of medication nonadherence.

DETAILED DESCRIPTION:
We will evaluate a dual component family-based intervention for adolescents with ADHD to improve medication adherence (Supporting Teen Adherence and Responsibility; STAR). STAR pairs Motivational Interviewing with parent-teen behavioral contracting. In the proposed study, adolescents with ADHD and a history of chronic nonadherence to their ADHD medication will be randomly assigned to medication alone (medication as usual: MAU) or MAU+STAR. They will be treated for 6 months with a 12 month maintenance period and 12 month followup. All interventions will occur at the offices of participants primary care physicians.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD; currently prescribed an FDA-approved medication for ADHD, history of medication nonadherence (taking less than 60% of prescribed doses); full scale Intelligence Quotient >80, no current language delay and/or had no language delays before age 3.

Exclusion Criteria:

* active medical conditions that could be worsened by stimulants (seizures, arrhythmias, hypertension) unless patient has clearance from primary specialist taking care of existing condition, pregnancy, Bipolar Disorder, schizophrenia, and/or other psychotic disorders, and diagnosis of current substance abuse or dependence (except nicotine), current psychotropic medication for conditions other than ADHD.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University Center for Children and Families, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No enrolled participants were excluded from the study prior to assignment to groups.
Groups:
- Medication as Usual + STAR: Medication as typically prescribed with the addition of the psychosocial intervention to improve medication adherence
  Medication as usual + STAR (Supporting Teen Adherence and Responsibility): Physicians will prescribe medication and adolescents and their parents will receive 6 sessions of psychosocial treatment to improve adolescents' motivation to use medication and to develop parent/teen contracting with the goal of setting medication adherence goals.
Period: Overall Study
Arm/Group | Medication as Usual | Medication as Usual + STAR
Started | 3 | 4
Completed (This study was prematurely discontinued due to low enrollment.) | 0 | 0
Not Completed | 3 | 4
Not completed — Premature discontinuation of study | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Medication as Usual + STAR: Medication as typically prescribed with the addition of the psychosocial intervention to improve medication adherence
  Medication as usual + STAR: Physicians will prescribe medication and adolescents and their parents will receive 6 sessions of psychosocial treatment to improve adolescents' motivation to use medication and to develop parent/teen contracting with the goal of setting medication adherence goals.
- Total: Total of all reporting groups
Arm/Group | Medication as Usual | Medication as Usual + STAR | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.00 (0.00) | 15.75 (0.50) | 14.33 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Proportion of prescribed doses taken as measured by electronic monitoring devices.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: Past 30 day proportion adherence
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
Past 30 day proportion adherence | .667 (.141) | 1.000 (NA) — Only 1 participant was analyzed in this group. Thus, it is not possible to calculate a standard deviation.

2. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Parent Report: Inattention
Description: Scores represent the total number of adolescent inattention symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) endorsed by parent on this rating scale. Possible scores range from 0 to 9 with higher scores representing the presence of more symptoms of inattention.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | 3.50 (4.95) | 7.00 (NA) — In this group, data are available for one participant only. Thus, it is not possible to calculate a standard deviation for this value.

3. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Parent Report: Hyperactive-Impulsive
Description: Scores represent the total number of adolescent hyperactive-impulsive symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) endorsed by parent on this rating scale. Possible scores range from 0 to 9 with higher scores representing the presence of more symptoms of hyperactivity-impulsivity.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | 1.00 (1.41) | 3.00 (NA) — In this group, data are available for 1 participant only. Thus, it is not possible to compute a standard deviation.

4. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Parent Report: Oppositional Defiant Disorder (ODD) Symptoms
Description: Scores represent the total number of adolescent symptoms of oppositional defiant disorder (ODD) endorsed by parent on this rating scale. Possible scores range from 0 to 8 with higher scores representing the presence of more symptoms of ODD.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | .50 (.71) | 0.00 (NA) — In this group, data are available for 1 participant only. Thus, it is not possible to compute a standard deviation.

5. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Parent Report: Conduct Disorder Symptoms
Description: Scores represent the total number of adolescent symptoms of conduct disorder (CD) endorsed by parent on this rating scale. Possible scores range from 0 to 15 with higher scores representing the presence of more symptoms of conduct disorder.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | .50 (.71) | 0.00 (NA) — In this group, data are available for 1 participant only. Thus, it is not possible to compute a standard deviation.

6. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Adolescent Report
Description: Scores represent the total number of self-reported adolescent inattention symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) endorsed on this rating scale. Possible scores range from 0 to 9 with higher scores representing the presence of more symptoms of inattention.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | 1.00 (1.41) | 0.00 (NA) — In this group, data are available for 1 participant only. Thus, it is not possible to compute a standard deviation.

7. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Adolescent Report: Hyperactive-Impulsive Symptoms
Description: Scores represent the total number of adolescent self-reported hyperactive-impulsive symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) endorsed on this rating scale. Possible scores range from 0 to 9 with higher scores representing the presence of more symptoms of hyperactivity-impulsivity.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | .50 (.71) | 0.00 (NA) — In this group, data are available for 1 participant only. Thus, it is not possible to compute a standard deviation.

8. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Adolescent Report: Oppositional Defiant Disorder Symptoms
Description: Scores represent the total number of adolescent self-reported symptoms of oppositional defiant disorder (ODD) symptoms endorsed on this rating scale. Possible scores range from 0 to 8 with higher scores indicating the presence of more symptoms of ODD.
Time Frame: Posttreatment (6 months)
Measure: Number; unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 1 | 1
score on a scale | 0 | 0

9. Secondary Outcome: Disruptive Behavior Disorder Rating Scale - Adolescent Report: Conduct Disorder Symptoms
Description: Scores represent the total number of self-reported adolescent symptoms of conduct disorder (CD) endorsed on this rating scale. Scores range from 0 to 15 with higher scores indicating the presence of more symptoms of CD.
Time Frame: Posttreatment (6 months)
Measure: Number; unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 1 | 1
score on a scale | 0 | 0

10. Secondary Outcome: Impairment Rating Scale - Parent Report
Description: Scores represent the average parent rating of adolescent functional impairment across multiple domains of functioning (i.e., home, school, peer relationships). Possible scores range from 0 to 6 with higher scores indicating more severe impairment and need for treatment.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | 2.58 (.82) | 2.17 (NA) — In this group, data are available for 1 participant only. Thus, it is not possible to compute a standard deviation.

11. Secondary Outcome: Impairment Rating Scale - Adolescent Report
Description: Scores represent the average adolescent self-report rating of adolescent functional impairment across multiple domains of functioning (i.e., home, school, peer relationships). Possible scores range from 0 to 6 with higher scores indicating more severe impairment and need for treatment.
Time Frame: Posttreatment (6 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 2 | 1
score on a scale | 1.42 (1.30) | .00 (NA) — In this group, data are available for 1 participant only. Thus, it is not possible to compute a standard deviation.

12. Secondary Outcome: Maintenance of Medication Adherence
Description: Continued monitoring of prescribed doses taken over 12-month monitoring period
Time Frame: 18 months
Population: Data were not collected.
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Followup Medication Adherence
Description: Continued monitoring of prescribed doses taken over 12-month followup period
Time Frame: 30 months
Population: Data were not collected.
Arm/Group | Medication as Usual | Medication as Usual + STAR
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Medication as Usual | Medication as Usual + STAR
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
Due to early termination of this study, only 3 participants (1 in the MAU+STAR arm and 2 in the MAU arm) reached the 6-month assessment. As a result, data should not be interpreted as indication of treatment effect due to the small sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No